CLINICAL TRIAL: NCT01246271
Title: a Retrospective Cohort Recognize the Out Comes of SUS With or Without Anterior Vaginal Repair
Brief Title: Sub Urethral Sling With or With Out Anterior Repair
Status: Completed | Type: Observational
Sponsor: Tabriz University (Other)
Responsible Party: Fatemeh Sadeghi Ghyassi, Iranian Center for EBM
Other Study IDs: 89-234; 8948 (Other: Tabriz University of Medical Sciences)
Record Dates: First submitted 2010-11-19; First posted 2010-11-23 (Estimated); Last update posted 2010-11-23 (Estimated); Status verified 2008-01

CONDITIONS: Urinary Incontinence
MeSH Terms: conditions — Urinary Incontinence

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Sub urethral sling
- sus with anterior vainal wall repair

SUMMARY:
There is a concern about choosing adequate surgical options for stress urinary incontinence associated with vaginal prolapsed and still lack of evidence can be observed. In this study we compared primary and secondary outcomes of single or combine surgery for SUI with pelvic organ prolapsed.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must be female
2. Subjective evidence of stress predominant symptoms on symptom specific questionnaire
3. Stress incontinence on urodynamics
4. Patients must be capable of filling in the symptom diary
5. Prolapse beyond the introitus

Exclusion Criteria:

1. Patients who are medically unfit to undergo surgical intervention.
2. Patients who have undergone previous continence surgery
3. Patients with voiding dysfunction
4. Patients with recurrent urinary tract infection
5. Patients who are not sure that their family is complete

Ages: 27 Years to 78 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: woman with stress urinary incontinence
Sampling Method: Probability Sample
Enrollment: 98 (Actual)
Dates: Start 2008-02; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Urinary incontinence cure rate according ICIQ-UIsf | 3 month after surgery

SECONDARY OUTCOMES:
morbidity and complication | 3 month after surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Urology department Imam Reza Hospital, Tabriz, Iran